CLINICAL TRIAL: NCT02546037
Title: Pilot Study to Determine the Effect of Different Dialyzer Membranes on Clotting During Haemodiafiltration Treatments in Patients With Chronic Kidney Disease
Brief Title: Clotting With Different Dialyzer Membranes
Acronym: TAGPSOLACEA
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: REC: 08/H0724/11
Record Dates: First submitted 2015-08-11; First posted 2015-09-10 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Kidney Failure
Keywords: coagulation; haemodialysis
MeSH Terms: conditions — Renal Insufficiency; Thrombosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SOLACEA 21H: single haemodiafiltration treatment using a SOLACEA 21H dialyzer (Nipro Corp, Osaka, Japan)
  Interventions: Device: SOLACEA 21H
- FX100: single haemodiafiltration treatment using a FX100 dialyzer (Fresenius MC, Bad Homburg, Germany)
  Interventions: Device: FX100 dialyzer

INTERVENTIONS:
Device: FX100 dialyzer — comparison of dialyzers
  Other Names: Fresenius FX 100
  Groups: FX100
Device: SOLACEA 21H — comparison of dialyzers
  Groups: SOLACEA 21H

SUMMARY:
Primary Objective:

The purpose of this study is to measure the amount of convection achieved with two different haemodiafilters designed for haemodiafiltration and clotting during haemodiafiltration treatment.

DETAILED DESCRIPTION:
This is a prospective observational cohort pilot study of patients under the care of the Royal Free Hospital with chronic kidney disease who have been established on regular thrice weekly haemodiafiltration treatments in a dialysis centre. Information on the study will be disseminated to the Royal Free consultant nephrologists at the dialysis centre with primary responsibility for the individual patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 years and older up to 80 years
* Under the care of the Royal Free Hospital with chronic kidney disease and established on regular thrice weekly haemodiafiltration.
* Able to provide written informed consent obtained

Exclusion Criteria:

* Patients scheduled for a kidney transplant
* Patients taking concomitant systemic anticoagulants
* Patients with known prothrombotic or bleeding disorders
* Patients with abnormal platelet counts
* Patients unable to provide written informed consent
* Patients not fulfilling inclusion criteria

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: attending RFH kidney care centre for routine outpatient HDF treatments for chronic kidney disease
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
convective volume exchanged | day 1
  volume of convective exchange achieved during the HDF session

SECONDARY OUTCOMES:
platelet and coagulation pathway activation | day 1
  measurement of coagulation pathway proteins and platelet activation markers
visual coagulation | day 1
  visual analogue score assessment of clotting in the extracorporeal circuit
small and middle sized solute clearances | day 1
  dialyzer clearance of small and middle sized molecules, including urea and beta 2 microglobulin

CONTACTS AND LOCATIONS:
Overall Officials: andrew davenport, Principal Investigator — UCL centre for nephrology, Royal Free Hospital